CLINICAL TRIAL: NCT06225622
Title: Dose Escalation and Expansion Clinical Trial of Irinotecan Liposome Combined With Oxaliplatin and 5-FU/LV Plus Bevacizumab as First-line Treatment of Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tianshu Liu, Head of Medical oncology, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K01
Record Dates: First submitted 2024-01-15; First posted 2024-01-26 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irinotecan liposome injection combined with oxaliplatin +5-FU/LV+ bevacizumab or cetuximab (Experimental): In dose escalation study, patients will be treated with irinotecan liposome injection combined with oxaliplatin +5-FU/LV+ bevacizumab. In expansion study, patients will be treated with irinotecan liposome injection combined with oxaliplatin +5-FU/LV+ bevacizumab or cetuximab, depending on their baseline mutation status. Oxaliplatin is accepted up to 12 cycles.
  Interventions: Drug: Irinotecan Liposome; Drug: Oxaliplatin; Drug: 5-FU; Drug: LV; Drug: Bevacizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Irinotecan Liposome — In dose escalation study, irinotecan liposome injection will be administered by an intravenous infusion at three doses of 60 mg/m2, 70 mg/m2 and 80 mg/m2, d1, 14 days per cycle. In expansion study, irinotecan liposome injection will be administered by an intravenous infusion at the dose of RP2D, d1, 14 days per cycle.
  Until the disease progresses or surgery is possible.
Drug: Oxaliplatin — 85 mg/m2, intravenously infusion, d1, 14 days per cycle, up to 12 cycles.
Drug: 5-FU — 2400mg/m2, intravenous infusion, d1-2, 14 days per cycle. Until the disease progresses or surgery is possible.
Drug: LV — 400mg/m2, intravenous infusion, d1, 14 days per cycle. Until the disease progresses or surgery is possible.
Drug: Bevacizumab — 5mg/kg, intravenous infusion, d1, 14 days per cycle. Until the disease progresses or surgery is possible.It is used to patients in dose escalation phase and with gene mutation in extension phase.
Drug: Cetuximab — 500mg/m2, intravenous infusion, d1, 14 days per cycle. Until the disease progresses or surgery is possible.For wild-type patients in extended phase studies.

SUMMARY:
Dose escalation clinical trial: To explore the dose limiting toxicity (DLT) of irinotecan liposome injection combined with oxaliplatin +5-FU/LV+ bevacizumab in first-line treatment of patients with advanced metastatic colorectal cancer, and to estimate the maximum tolerated dose (MTD) of combined administration.

Expansion clinical trial: To evaluate the safety and efficacy of irinotecan liposome injection combined with oxaliplatin +5-FU/LV+ bevacizumab or cetuximab in first-line treatment of patients with advanced metastatic colorectal cancer. Exploratory analysis of ctDNA changes and genetic mutations in patients at baseline.

DETAILED DESCRIPTION:
This is a dose escalation and expansion study to evaluate the safety and efficacy of irinotecan liposome injection in patients with first-line treatment for metastatic colorectal cancer. In the dose escalation phase, patients will be treated with a combination regimen of irinotecan liposome injection at doses of 60mg/m2, 70mg/m2, and 80mg/m2, and 9 to 18 eligible patients are expected to be enrolled. In the expansion phase, approximately 60 patients will receive combination therapy with irinotecan liposome RP2D dose and exploratory analysis of genetic mutations at baseline and ctDNA changes during treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old.
* Histopathologically confirmed patient with an inoperable metastatic colorectal adenocarcinoma.
* The unresectable stage of metastatic disease has not received any systemic antitumor therapy.
* For subjects previously receiving neoadjuvant or adjuvant therapy, the date of first discovery of disease progression must be at least 12 months removed from the date of last administration of neoadjuvant or adjuvant therapy.
* The presence of at least 1 measurable lesion that can be evaluated according to the RECIST v1.1 criteria.
* ECOG 0
* Normal bone marrow and organ function: ① Neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥100×10^9/L, hemoglobin (Hb) ≥90g/L, white blood cells (WBC) ≥3.0×10^9/L, albumin (ALB) ≥35 g/L, and no bleeding tendency; ② AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred; The total bilirubin level doesn't exceed the upper limit of the agency's normal range; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockroft-Gault)
* Understand the situation of this study, patients and/or legal representatives voluntarily agree to participate in this study and sign informed consent form.

Exclusion Criteria:

* Patients with known MSI-H or dMMR who were evaluated by investigators as suitable for treatment with immune checkpoint inhibitors.
* Patients allergic to the investigational drug and its excipients.
* Underweight (body mass index [BMI]<18.5 kg/m^2).
* Known or suspected central nervous system metastasis.
* Received irinotecan before enrollment.
* Had undergone surgery and other oncologic treatments within the first 4 weeks of enrollment.
* Previous treatment-related toxicity didn't return to NCI-CTCAE v5.0 class I or below.
* The use of CYP3A, CYP2C8, and UGT1A1 inhibitors or inducers couldn't be discontinued or were not discontinued within 2 weeks prior to enrollment.
* Serious gastrointestinal disorders.
* Interstitial lung disease.
* Tendency of arterial embolism and massive bleeding within 6 months before enrollment (except surgical bleeding).
* Patients with fluid accumulation that couldn't reach a stable state and small amount of pleural effusion or ascites on imaging without clinical symptoms could be enrolled.
* Intestinal obstruction, signs and symptoms of intestinal obstruction, or the stent has been previously implanted and the stent has not been removed before the screening period.
* Gastrointestinal perforation, intraperitoneal abscess, and fistula.
* Any serious or uncontrolled systemic disease, including uncontrolled high blood pressure, heart disease, active bleeding, active viral infection, etc.
* Have had other malignancies within the past 5 years or currently, except cured cervical carcinoma in situ, uterine carcinoma in situ, and non-melanoma skin cancer.
* Patients of childbearing age who refuse to take contraceptives, women who are pregnant or breastfeeding.
* The researchers didn't consider it appropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose | Up to 14 days
  To investigate the safety.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Start by signing the informed consent form until 4 weeks after the last dose.
  To evaluate the incidence and severity of hematological adverse events in patients.

SECONDARY OUTCOMES:
Objective response rate | From initial medication to the date of first documented progression or end of medication, assessed up to 20 months.
  To investigate the preliminary antitumor efficacy of study.
Disease control rate | From initial medication to the date of first documented progression or end of medication , assessed up to 20 months.
  To investigate the preliminary antitumor efficacy of study.
Progression free survival | From initial medication to the date of first documented progression or date of death from any cause, whichever came first , assessed up to 22 months.
  To investigate the preliminary antitumor efficacy of study.
R0 resection | From the first dose to the surgery, assessed up to 22 months.
  To assess surgical conversion rates in patients who could be surgically resected.

OTHER OUTCOMES:
Changes of tumor ctDNA | From initial medication to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  To investigate the preliminary antitumor effect of this study and the relationship between ctDNA changes and disease prognosis.
Gene polymorphism | Within a month of enrollment.
  To investigate the polymorphism of UGT1A1 and colorectal cancer genes at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China